CLINICAL TRIAL: NCT04446468
Title: Prevention of Suicide in Veterans Through Brief Intervention and Contact (VA-BIC)
Brief Title: Suicide Prevention Study of VA-BIC in the Veteran Population
Acronym: VA-BIC RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MHBC-007-19F
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Suicide Prevention
Keywords: Mental health education; Clinical Trial; Suicidal ideation; Suicide, attempted
MeSH Terms: conditions — Suicide Prevention; Suicidal Ideation; Suicide, Attempted | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel: PEACE plus standard psychiatric discharge care vs. standard psychiatric discharge care alone
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to treatment allocation and will remind the participant at each contact to not disclose their treatment status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEACE (Experimental): The PEACE intervention will be delivered by a trained mental health staff member, such as a study psychologist, mental health nurse, social worker, or psychiatrist. The intervention consists of three synergistic components that work to support the patient after inpatient psychiatric discharge: 1) Brief educational component, where the patient receives a one-hour, one-on-one, personalized educational session on suicide prevention; 2) Seven regular contacts after discharge, where the study psychologist who delivered the brief educational visit will contact the patient to monitor the patient's symptoms, assess treatment adherence, review their safety plan, and assist the patient with engaging in care, if needed; and 3) Mobile app, which aims to improve the patient's social connectedness and provide additional educational materials on suicide. Patients in this arm will also continue to receive standard post-discharge psychiatric care.
  Interventions: Behavioral: PEACE; Other: Standard Psychiatric Hospital Discharge Care
- Control (Experimental): Those randomized to the control arm will receive standard psychiatric hospital discharge care alone. Current VA standard discharge care includes five core elements. First, patients and their outpatient providers are required to be involved in discharge planning. Second, patients should be offered evidence-based treatments to address their mental health symptoms. Third, the inpatient team should work with the patient to complete a safety plan prior to discharge. Fourth, the inpatient team should arrange two follow-up care visits within 30 days of discharge. Fifth, the inpatient team in conjunction with the SPC assess whether patients are appropriate to be placed on the High Risk for Suicide List. Patients who are placed on the High Risk for Suicide List receive enhanced oversight as outlined in VA policy.
  Interventions: Other: Standard Psychiatric Hospital Discharge Care

INTERVENTIONS:
Behavioral: PEACE — The intervention consists of three synergistic components that work to support the patient after inpatient psychiatric discharge: 1) Brief educational component, where the patient receives a one-hour, one-on-one, personalized educational session on suicide prevention; 2) Seven regular contacts after discharge, where the study psychologist who delivered the brief educational visit will contact the patient to monitor the patient's symptoms, assess treatment adherence, review their safety plan, and assist the patient with engaging in care, if needed; and 3) Mobile app, which aims to improve the patient's social connectedness and provide additional educational materials on suicide.
  Arms: PEACE
Other: Standard Psychiatric Hospital Discharge Care — Current VA standard discharge care includes five core elements. First, patients and their outpatient providers are required to be involved in discharge planning. Second, patients should be offered evidence-based treatments to address their mental health symptoms. Third, the inpatient team should work with the patient to complete a safety plan prior to discharge. Fourth, the inpatient team should arrange two follow-up care visits within 30 days of discharge. Fifth, the inpatient team in conjunction with the SPC assess whether patients are appropriate to be placed on the High Risk for Suicide List. Patients who are placed on the High Risk for Suicide List receive enhanced oversight as outlined in VA policy.
  Other Names: Standard Care

SUMMARY:
The VA is committed to reducing suicide in the U.S. Veteran population. Over 6,000 Veterans die from suicide each year, and this risk is particularly high following a psychiatric hospitalization. This may be due to problems with engagement in care and poor social connectedness. Although the VA has implemented tools to address Veteran suicide risk, suicide after psychiatric discharge remains an ongoing problem. This has highlighted the need to develop new interventions and approaches to post-discharge mental health care within the VA. In response, this project is a randomized control trial of an intervention an intervention called Prevention of suicide: Education, Awareness, Connection, and Engagement (PEACE). This intervention is comprised of two synergistic and promising components to prevent suicide: 1) a mobile mental health app, which aims to improve social connectedness after discharge; and 2) a manual-based intervention called the Veterans Affairs Brief Intervention and Contact Program (VA-BIC), which promotes engagement in care. The overall goal of this study is to determine if the PEACE intervention combined with standard discharge care reduces suicidal ideation as compared to a control group receiving only standard discharge care.

DETAILED DESCRIPTION:
Background: Suicide is a major public health concern in the U.S., and even more so in the Veteran population. Furthermore, the period following psychiatric hospitalization is one of the highest risk periods for suicide. Based on current evidence, some of the most important contributing factors to post-hospitalization suicide risk include problems with engagement in care, fragmented care, and lack of social connectedness. Other studies in civilian populations have also raised similar concerns, highlighting the need to identify novel and effective interventions or approaches to post-discharge mental health care.

Objectives: This project aims to 1) Identify the effect of PEACE on suicidal ideation after psychiatric hospitalization, compared to standard care alone; 2) Identify the effect of PEACE on social connectedness and engagement in care after psychiatric hospitalization, compared to standard care alone; and 3) Compare the effect of PEACE on suicide attempts and suicide deaths after psychiatric hospitalization, compared to standard care alone.

Methods: This is a single-site, assessor-blinded, randomized control trial of PEACE plus standard psychiatric hospital discharge care compared to standard psychiatric hospital discharge care alone. The trial will enroll up to 160 participants aged 18 years and older who are being discharged from the White River Junction VA Medical Center inpatient mental health unit. Participants will be randomized to either the PEACE intervention plus standard psychiatric discharge care or standard psychiatric discharge care alone. Suicidal ideation, hopelessness, social connectedness, engagement in care, suicide attempts, and app engagement (only those randomized to PEACE) will be measured at baseline and one, three, and six months post-discharge. Participants randomized to PEACE will also receive eight additional intervention contacts as part of the VA-BIC protocol.

Hypothesis: Veterans receiving the PEACE intervention will report greater improvements in suicidal thoughts and behaviors, hopelessness, social connectedness, and engagement in care at follow-up contact visits compared to Veterans receiving standard care alone.

ELIGIBILITY:
Inclusion Criteria:

* Per the unit psychiatrist, hospitalization was due to concerns about acute risk for self-harm including suicidal ideation, suicide attempt, and/or admitting provider deemed the patient was at imminent risk for self-harm;
* Be a Veteran eligible to receive VA services;
* Be 18 years or older;
* Be able to speak English;
* Have access to a smart phone and express willingness to download a mobile app.

Exclusion Criteria:

* Unable to provide informed consent;
* The investigators do not plan to enroll any potentially vulnerable populations including prisoners, or involuntarily committed patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Riblet, MD MPH, Principal Investigator — White River Junction VA Medical Center, White River Junction, VT
Locations (1):
- White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cornelius SL, Berry T, Goodrich AJ, Shiner B, Riblet NB. The Effect of Meteorological, Pollution, and Geographic Exposures on Death by Suicide: A Scoping Review. Int J Environ Res Public Health. 2021 Jul 23;18(15):7809. doi: 10.3390/ijerph18157809. PMID 34360101
- [Background] Riblet NB, Gottlieb DJ, Watts BV, Levis M, Shiner B. Irregular hospital discharge from acute inpatient and residential mental health treatment settings in a large integrated healthcare system. Gen Hosp Psychiatry. 2021 Sep-Oct;72:7-14. doi: 10.1016/j.genhosppsych.2021.06.009. Epub 2021 Jun 26. PMID 34214935
- [Background] Riblet NB, Gottlieb DJ, Watts BV, Levis M, Scott R, Shiner B. Is It Time for the Mental Health Field to Consider Unplanned Discharge a Key Metric of Patient Safety? J Nerv Ment Dis. 2022 Mar 1;210(3):227-230. doi: 10.1097/NMD.0000000000001425. PMID 35199662
- [Background] Riblet NB, Kenneally L, Stevens S, Watts BV, Gui J, Forehand J, Cornelius S, Rousseau GS, Schwartz JC, Shiner B. A virtual, pilot randomized trial of a brief intervention to prevent suicide in an integrated healthcare setting. Gen Hosp Psychiatry. 2022 Mar-Apr;75:68-74. doi: 10.1016/j.genhosppsych.2022.02.002. Epub 2022 Feb 18. PMID 35202942
- [Background] Riblet NB, Varela M, Ashby W, Zubkoff L, Shiner B, Pogue J, Stevens SP, Wasserman D, Watts BV. Spreading a Strategy to Prevent Suicide After Psychiatric Hospitalization: Results of a Quality Improvement Spread Initiative. Jt Comm J Qual Patient Saf. 2022 Oct;48(10):503-512. doi: 10.1016/j.jcjq.2022.02.009. Epub 2022 Mar 6. PMID 35382976
- [Background] Britton PC, Berrouiguet S, Riblet NB, Zhong BL. Editorial: Brief interventions in suicide prevention across the continuum of care. Front Psychiatry. 2022 Jul 26;13:976855. doi: 10.3389/fpsyt.2022.976855. eCollection 2022. No abstract available. PMID 35958652
- [Background] Riblet NB, Matsunaga S, Lee Y, Young-Xu Y, Shiner B, Schnurr PP, Levis M, Watts BV. Tools to Detect Risk of Death by Suicide: A Systematic Review and Meta-Analysis. J Clin Psychiatry. 2022 Nov 16;84(1):21r14385. doi: 10.4088/JCP.21r14385. PMID 36383739
- [Background] Riblet NB, Shiner B, Young-Xu Y, Watts BV. Lithium in the prevention of suicide in adults: systematic review and meta-analysis of clinical trials. BJPsych Open. 2022 Nov 17;8(6):e199. doi: 10.1192/bjo.2022.605. PMID 36384820
- [Background] Riblet NB, Matsunaga S, Shiner B, Schnurr PP, Watts BV. Are suicide risk scales sensitive to change? A scoping review. J Psychiatr Res. 2023 May;161:170-178. doi: 10.1016/j.jpsychires.2023.03.007. Epub 2023 Mar 9. PMID 36931135
- [Background] Riblet NBV, Watts BV. Another Reason to Quit Smoking: Results of a Prospective Study Examining Smoking, COPD, and Suicide. Chest. 2023 Feb;163(2):259-261. doi: 10.1016/j.chest.2022.10.016. No abstract available. PMID 36759108
- [Background] Riblet NB, Young-Xu Y, Shiner B, Schnurr PP, Watts BV. The efficacy and safety of buprenorphine for the treatment of depression: A systematic review and meta-analysis. J Psychiatr Res. 2023 May;161:393-401. doi: 10.1016/j.jpsychires.2023.03.037. Epub 2023 Mar 30. PMID 37019069
- [Background] Riblet NB, Soncrant C, Mills P, Yackel EE. Analysis of Reported Suicide Safety Events Among Veterans Who Received Treatment Through Department of Veterans Affairs-Contracted Community Care. Mil Med. 2023 Aug 29;188(9-10):e3173-e3181. doi: 10.1093/milmed/usad088. PMID 37002596
- [Background] Riblet NB, Gottlieb DJ, Shiner B, Zubkoff L, Rice K, Watts BV, Rusch B. An Analysis of Irregular Discharges From Residential Treatment Programs in the Department of Veterans Affairs Health Care System. Mil Med. 2023 Nov 3;188(11-12):e3657-e3666. doi: 10.1093/milmed/usad131. PMID 37167031
- [Background] Kenneally L, Stevens S, Cornelius S, Shiner B, Rice K, Park J, Watts BV, Teja N, Riblet N. Pilot randomized controlled trial of a brief strategy to prevent suicide after discharge from residential addiction treatment. J Subst Use Addict Treat. 2023 Nov;154:209156. doi: 10.1016/j.josat.2023.209156. Epub 2023 Aug 29. PMID 37652208

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PEACE | Control
Started | 46 | 46
Completed | 33 | 35
Not Completed | 13 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEACE | Control | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.33 (15.66) | 46.52 (13.93) | 48.42 (14.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 14
  Male | 42 | 36 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 43 | 40 | 83
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 44 | 43 | 87
  Unknown or Not Reported | 0 | 0 | 0
Beck Scale for Suicide Ideation (BSS) [Mean (Standard Deviation); unit: units on a scale] — The BSS is a self-reported questionnaire that assesses severity of suicidal ideation. BSS scores range from 0-38. While no established cutoff score exists to delineate risk of suicide, higher scores indicate more severe suicidal ideation. Scores were calculated at baseline.
  units on a scale | 13.80 (10.75) | 13.59 (9.44) | 13.70 (10.06)
The Beck Scale for Hopelessness (BHS) [Mean (Standard Deviation); unit: units on a scale] — The BHS measures hopelessness and scores range from 0-20 with higher scores reflecting worse hopelessness. BHS scores were calculated at baseline.
  units on a scale | 10.72 (6.31) | 11.04 (5.79) | 10.88 (6.02)
Partners in Health Scale (PIH): Self-Management [Mean (Standard Deviation); unit: units on a scale] — The PIH measures self-management of their chronic health conditions. Scores range from 0-96 with higher scores indicated greater self-management and engagement. PIH scores were calculated at baseline.
  units on a scale | 60.83 (15.42) | 59.89 (13.26) | 60.36 (14.31)
Interpersonal Needs Questionnaire-15 (INQ-15), perceived burdensomeness [Mean (Standard Deviation); unit: units on a scale] — The INQ-15 is a 15 item scale that measures thwarted belongingness and perceived burdensomeness. Each item is measured on a 7-point Likert scale. Items 7, 8, 10, 13, 14, and 15 are reverse coded. Scores on the total scale range from 15-105. The perceived burdensomeness subscale includes 6 items and scores range from 6-42 with higher scores indicating worse perceived burdensomeness. Perceived burdensomeness scores were calculated at baseline.
  units on a scale | 20.61 (10.58) | 20.30 (10.50) | 20.46 (10.48)
Interpersonal Needs Questionnaire-15 (INQ-15), thwarted belongingness [Mean (Standard Deviation); unit: units on a scale] — The INQ-15 is a 15 item scale that measures thwarted belongingness and perceived burdensomeness. Each item is measured on a 7-point Likert scale. Items 7, 8, 10, 13, 14, and 15 are reverse coded. Scores on the total scale range from 15-105. The thwarted belongingness subscale includes 9 items and scores range from 9-63 with higher scores indicating worse thwarted belongingness. Thwarted belongingness scores were calculated at baseline.
  units on a scale | 39.52 (11.40) | 38.04 (12.42) | 38.78 (11.87)
The Multidimensional Scale of Perceived Social Support (MSPSS) [Mean (Standard Deviation); unit: units on a scale] — The MSPSS is a 12-item valid scale that assesses perceived support from family, friends and significant others. The scores on the scale range from 1-7 with higher scores suggesting greater perceived support. MSPSS scores were measured at baseline.
  units on a scale | 4.16 (1.68) | 4.51 (1.52) | 4.33 (1.60)
Suicide Related Coping Scale (SRCS) [Mean (Standard Deviation); unit: units on a scale] — The SRCS is a valid scale that includes 17 items that measure a patient's perception of their ability to cope with suicidal thoughts and behaviors. The scale includes a subscale that reports on external coping as well as another subscale that reports on internal coping. The total scores on the SRCS range from 0-68 with higher scores suggesting greater ability to cope with suicidal ideation and behavior. SRCS scores were measured at baseline.
  units on a scale | 44.30 (12.62) | 46.48 (11.18) | 45.39 (11.90)
MINI International Neuropsychiatric Interview: Current mental health conditions [Mean (Standard Deviation); unit: sum of mental health conditions] — The MINI International Neuropsychiatric Interview is a short, structured diagnostic interview that has been validated against the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders. The MINI was used to assess the sum of current mental health conditions that were present at baseline.
  sum of mental health conditions | 2.9 (0.9) | 2.6 (0.9) | 2.73 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Beck Scale for Suicide Ideation (BSS)
Description: The BSS is a self-reported questionnaire that assesses severity of suicidal ideation. The BSS measures attitudes, behaviors, and plans to die by suicide. Each item on the BSS is scored on a scale from 0 to 2 and the first 19 of the 21 items are used to calculate a total score ranging from 0 - 38. The BSS has high reliability and is a valid measure of suicidal ideation. There is also evidence that the BSS is measurement invariant across time. The BSS is widely used in clinical trials, is sensitive to clinical change, and unlike most other measures of suicidal ideation, higher scores on the BSS are associated with death by suicide. While there is no established BSS cutoff score to classify suicide risk as high, low, or none, there is evidence that higher scores on the BSS correspond to more severe suicidal ideation.
Time Frame: 1-month, 3-month, and 6- month post-discharge
Population: The number analyzed differs across follow-up periods due to loss to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PEACE | Control
Number analyzed (Participants) | 36 | 38
units on a scale
  1 month post discharge | 7.8 (8.75) | 7.61 (9.13)
  3 month post discharge: number analyzed (Participants) | 34 | 36
  3 month post discharge | 9.21 (8.64) | 6.78 (8.49)
  6 month post discharge: number analyzed (Participants) | 33 | 34
  6 month post discharge | 8.03 (9.88) | 5.71 (8.78)

2. Secondary Outcome: Suicide-Related Coping Scale (SRCS)
Description: This scale includes 17 questions related to a patient's perception of their ability to cope with suicidal thoughts. Each item is assessed using a 5-point Likert scale and the measure has been developed based on two studies of suicide prevention strategies conducted within Veteran populations. The scale includes two subscales including an External Coping subscale and an Internal Coping Subscale. Both subscales have shown good acceptable internal consistency. The two factors are also sensitive to change over time. The score range for the entire scale is 0-68. Higher scores on the scale suggest better coping.
Time Frame: 1-month, 3-month, and 6- month post-discharge
Population: The number analyzed differs across follow-up periods due to loss to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PEACE | Control
Number analyzed (Participants) | 36 | 38
units on a scale
  1 month post discharge | 52.86 (9.82) | 53.21 (9.88)
  3 months post discharge: number analyzed (Participants) | 34 | 36
  3 months post discharge | 52.47 (9.33) | 53.39 (11.16)
  6 months post discharge: number analyzed (Participants) | 33 | 32
  6 months post discharge | 52.94 (11.82) | 56.44 (10.25)

3. Secondary Outcome: The Partners in Health Scale (PIH): Self-Management
Description: The Partners in Health Scale measures self-management of chronic health conditions. It is a valid scale that includes 12 items. Each question is measured on a Likert scale of 0-8. Scores range from 0-96. Higher scores reflect improved engagement and self-management of chronic health conditions.
Time Frame: 1-month, 3-months, and 6-months post discharge
Population: The number analyzed differs across follow-up periods due to loss to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PEACE | Control
Number analyzed (Participants) | 36 | 38
units on a scale
  1 month post discharge | 73.25 (14.70) | 73.29 (12.27)
  3 months post discharge: number analyzed (Participants) | 34 | 36
  3 months post discharge | 71.0 (14.34) | 73.19 (12.03)
  6 months post discharge: number analyzed (Participants) | 33 | 32
  6 months post discharge | 73.97 (12.71) | 75.94 (12.55)

4. Secondary Outcome: Beck Hopelessness Scale (BHS)
Description: The BHS is a 20-item self-report scale that assesses hopelessness over the past seven days. Patients comment on feelings about the future, loss of motivation, and future expectations. Total scores range from 0 to 20, with higher scores suggesting more hopelessness. Higher scores on the BHS are associated with increased suicide risk. The BHS has good reliability and validity and is sensitive to change.
Time Frame: 1-month, 3-months and 6- months post-discharge
Population: The number analyzed differs across follow-up periods due to loss to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PEACE | Control
Number analyzed (Participants) | 36 | 38
units on a scale
  1 month post discharge | 8.19 (5.96) | 7.66 (6.19)
  3 months post discharge: number analyzed (Participants) | 34 | 37
  3 months post discharge | 9.0 (6.0) | 6.57 (5.06)
  6 months post discharge: number analyzed (Participants) | 33 | 35
  6 months post discharge | 8.0 (5.65) | 5.57 (5.22)

5. Secondary Outcome: Interpersonal Needs Questionnaire-15 (INQ-15): Thwarted Belongingness
Description: The INQ-15 is a 15 item scale that measures thwarted belongingness and perceived burdensomeness. Each item is measured on a 7-point Likert scale. Items 7, 8, 10, 13, 14, and 15 are reverse coded. Scores on the total scale range from 15-105. The thwarted belongingness subscale includes 9 items and scores range from 9-63 with higher scores indicating worse thwarted belongingness.
Time Frame: 1 month, 3-months, and 6-months post discharge
Population: The number analyzed differs across follow-up periods due to loss to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PEACE | Control
Number analyzed (Participants) | 36 | 38
units on a scale
  1 month post discharge | 31.47 (12.64) | 28.45 (13.43)
  3 months post discharge: number analyzed (Participants) | 34 | 36
  3 months post discharge | 33.85 (14.07) | 30.81 (14.81)
  6 months post discharge: number analyzed (Participants) | 33 | 34
  6 months post discharge | 32.52 (13.56) | 25.79 (12.09)

6. Secondary Outcome: Interpersonal Needs Questionnaire-15 (INQ-15): Perceived Burdensomeness
Description: The INQ-15 is a 15 item scale that measures thwarted belongingness and perceived burdensomeness. Each item is measured on a 7-point Likert scale. Items 7, 8, 10, 13, 14, and 15 are reverse coded. Scores on the total scale range from 15-105. The perceived burdensomeness subscale includes 6 items and scores range from 6-42 with higher scores indicating worse perceived burdensomeness.
Time Frame: 1-month, 3-months, and 6-months post discharge
Population: The number analyzed differs across follow-up periods due to loss to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PEACE | Control
Number analyzed (Participants) | 36 | 38
units on a scale
  1 month post discharge | 15.03 (9.64) | 13.68 (8.82)
  3 months post discharge: number analyzed (Participants) | 34 | 37
  3 months post discharge | 14.53 (8.20) | 13.78 (8.82)
  6 months post discharge: number analyzed (Participants) | 33 | 34
  6 months post discharge | 13.18 (7.54) | 11.5 (8.15)

7. Secondary Outcome: The Multidimensional Scale of Perceived Social Support (MSPSS)
Description: The multidimensional scale of perceived social support is a valid scale that includes 12 items that measure several perceived sources of social support including family, friends, and significant others. The score range is 1-7 with higher scores suggesting greater perceived support.
Time Frame: 1-month, 3-months and 6- months post-discharge
Population: The number analyzed differs across follow-up periods due to loss to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PEACE | Control
Number analyzed (Participants) | 36 | 38
units on a scale
  1 month post discharge | 4.85 (1.57) | 5.16 (1.42)
  3 months post discharge: number analyzed (Participants) | 34 | 36
  3 months post discharge | 4.69 (1.70) | 4.66 (2.0)
  6 months post discharge: number analyzed (Participants) | 33 | 32
  6 months post discharge | 4.87 (1.59) | 5.33 (1.45)

8. Secondary Outcome: App Engagement Scale (AES) for Mobile Applications
Description: The App Engagement Scale (AES) is adapted from the Mobile Application Rating Scale (uMARS) and is a valid scale. All items are rated on a 5-point scale. Scores range from 0-40 and higher scores indicate greater perceived quality of the mobile application.
Time Frame: 6- month post-discharge
Population: The app that was planned to be used for this study was available in the public domain when designing the study, but became non-functional during the course of the study. Thus participants were unable to access the app. The participants therefore did not answer the questions on the AES scale because they could not comment on the quality of the mobile application as they did not access the app.
Arm/Group | PEACE | Control
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Continuity of Care
Description: There is some evidence that improved continuity of care may lead to better mental health outcomes. However, a single valid standardized measure of continuity of care for mental health has not been described in the literature. Continuity of care was measured by assessing the total number of VA outpatient mental health visits attended within the three months after discharge.
Time Frame: 3-months post discharge
Measure: Mean (Standard Deviation); unit: mental health visits attended
Arm/Group | PEACE | Control
Number analyzed (Participants) | 46 | 46
mental health visits attended | 14.32 (12.14) | 14.15 (10.31)

10. Secondary Outcome: Suicide Attempts: Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS includes a 7-item subscale that assesses for actual and interrupted suicide attempts. It is a valid and reliable scale that includes a seven-item subscale that asks patients to self-report on actual attempts, interrupted attempts, aborted attempts, and preparatory acts or behaviors. The C-SSRS subscale was used specifically to assess the number of participants who had an actual fatal or non-fatal suicide attempt within the first 6 months post discharge.
Time Frame: Baseline to 6- months post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | PEACE | Control
Number analyzed (Participants) | 46 | 46
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: Baseline to end of follow-up, up to 6 months.
Description: Because our study enrolled a high-risk group of patients, it was anticipated that patients would potentially report worsening mental health symptoms and/or problems specific to substance use. We expected that patients may experience suicidal behavior and related outcomes. In some cases, the patients would be expected to be hospitalized or treated in the emergency room for these reasons. Based on local approval from our institutional review board, we treated these events as adverse events.
Arm/Group | PEACE | Control
All-Cause Mortality (participants affected / at risk) | 2/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 1/46 | 0/46
Other Adverse Events (participants affected / at risk) | 18/46 | 15/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEACE (N=46) | Control (N=46)
death due to natural causes (General disorders) | 1 | 0 — the death was deemed to be due to natural causes by the state medical examiner
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEACE (N=46) | Control (N=46)
non-fatal or fatal suicide attempt (Psychiatric disorders) | 3 | 3
Suicidal behavior (preparatory or planning behaviors, interrupted attempt, or self-aborted attempt) (Psychiatric disorders) | 2 | 3
worsening mental health symptoms (Psychiatric disorders) | 14 | 11 — worsening mental health symptoms (e.g. anxiety) that were self-reported to study staff (either interventionist or assessor) during the course of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT04446468/Prot_SAP_001.pdf
  • Informed Consent Form (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT04446468/ICF_000.pdf